CLINICAL TRIAL: NCT02283879
Title: Human Umbilical Cord Mesenchymal Stem Cell Therapy for Patients With Cerebral Hemorrhage
Brief Title: Human Umbilical Cord Mesenchymal Stem Cell in Cerebral Hemorrhage Sequela
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shenzhen Hornetcorn Bio-technology Company, LTD (Industry)
Collaborators: Fifth Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYK-Cerebral hemorrhage
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2015-07

CONDITIONS: Cerebral Hemorrhage
Keywords: Human Umbilical Cord Mesenchymal Stem Cell; Mesenchymal Stem Cell; Cerebral hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hUC-MSC treatment (Experimental): Patients will receive human umbilical cord mesenchymal stem cells transplantation with a 12 months follow-up.
  Interventions: Biological: Human umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Human umbilical cord mesenchymal stem cells — A single dose of 2×107 hUC-MSC will treated to patients, IV, Repeat every weeks for four times.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of human umbilical cord mesenchymal stem cell(hUC-MSC) for cerebral hemorrhage sequela.

DETAILED DESCRIPTION:
Human umbilical cord mesenchymal stem cells exhibit the potential to differentiate into neural cells, which have been confirmed in in vivo and in vitro experiments. There have been few clinical reports describing umbilical cord mesenchymal stem cells for treatment of cerebral hemorrhage.

To investigate the effects of hUC-MSC treatment for cerebral hemorrhage sequela, 20 patients with cerebral hemorrhage will be enrolled and receive 4 times of hUC-MSC transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-70 intracerebral hemorrhage patient
* With stroke history of more than 3 months, less than 60 months
* National Institutes of Health stroke scale(NIHSS) score of 7 or more points
* Patient is stable (normal respiration, afebrile, BP less than mean arterial pressure of 125 mm of Hg, fasting blood sugar <7 mg, and normal urea/electrolytes for at least 48 hours.)

Exclusion Criteria:

* History of neurological disease, head injury or psychiatric disorder;
* Pregnant women;
* Impaired liver function, abnormal blood coagulation, AIDS, HIV, combine other tumor or special condition;
* Progressive apoplexy;
* With malignant tumors.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation through vital signs, the results of clinical lab tests and adverse events (AEs) | 12 months

SECONDARY OUTCOMES:
Improvement of infarct size measured by brain MRI | before the transplant and 1, 6, 12 months after transplantation
Modified Barthel index | before and 1, 3, 6 and 12 months after transplantation
National Institutes of Health stroke scale(NIHSS) score | before the transplant and after the transplant 1, 2 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ping J Chen, Professor, Principal Investigator — Fifth Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Fifth Affiliated Hospital Immunotherapy center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided